CLINICAL TRIAL: NCT06658509
Title: Regulation of Different Types of Interval Training on Vascular Function of Overweight Female University Students
Brief Title: Regulation of Different IT on Vascular Function of Overweight Female University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RODTOITOVFOOFUS
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Overweight
Keywords: High intensity interval training; Sprint interval training; Overweight; Female; Vascular function
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIIT group (Experimental)
  Interventions: Behavioral: HIIT
- SIT group (Experimental)
  Interventions: Behavioral: SIT
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: HIIT — High-intensity interval training
  Arms: HIIT group
Behavioral: SIT — Sprint interval training
  Arms: SIT group

SUMMARY:
This study investigates the effects of different interval training methods, specifically high-intensity interval training (HIIT) and sprint interval training (SIT), on vascular function in overweight female university students. A randomized controlled trial was conducted over an 8-week period.

DETAILED DESCRIPTION:
This study aimed to evaluate how different types of interval training (HIIT and SIT) influence vascular function in overweight female university students. Participants were initially enrolled and randomly assigned to HIIT, SIT, or control groups. The participants in HIIT and SIT groups underwent an 8-week supervised exercise program 3 times per week on a treadmill. Both pre- and post-intervention measurements were taken, including vascular function, morphological indicators, and blood markers. This study highlights the potential of interval training as a time-efficient and effective intervention for improving cardiovascular health and body composition in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 25 years, female.
* Participants' BMI more than 24 kg·m-2.
* Participants without regular exercise habits.

Exclusion Criteria:

* Participants underwent other interventions (e.g., nutrition, psychology, exercise, health education, et al).
* Participants had a history of systematic and professional exercise habit.
* Participants presenced of disease or condition restricting participation, such as injuries, respiratory disease or cardiovascular diseases.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Brachial-ankle pulse wave velocity (baPWV) | 8 weeks
  The change of baPWV before and after intervention.
Ankle-brachial index (ABI) | 8 weeks
  The change of ABI before and after intervention.
Nitric oxide (NO) | 8 weeks
  The change of NO before and after intervention.
Endothelin (ET) | 8 weeks
  The change of ET before and after intervention.
Body weight (BW) | 8 weeks
  The change of BW before and after intervention.
Body mass index (BMI) | 8 weeks
  The change of BMI before and after intervention.
Body fat% (BF%) | 8 weeks
  The change of BF% before and after intervention.

SECONDARY OUTCOMES:
Height | 8 weeks
  The change of height before and after intervention.
Blood pressure (BP) | 8 weeks
  The change of BP before and after intervention.
Maximal oxygen uptake (VO2max) | 8 weeks
  The change of VO2max before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: No